CLINICAL TRIAL: NCT07400874
Title: The Effects of Acupressure, Aromatherapy, and Virtual Reality on Pain, Fear, and Anxiety in Children During Blood Sampling Procedures
Brief Title: Use of Acupressure, Aromatherapy, and Virtual Reality for Children in During Blood Collection Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Gamze Akay, Assistant Professor, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Blood Collection and Child
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Blood Collection
Keywords: Blood Collection; Fear; Pain; Anxiety; Acupressure; Virtual reality; listening music; child
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine clinical care will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): Before blood is drawn, the child will undergo acupressure, watch a video through virtual reality glasses, and listen to music through headphones.
  Interventions: Other: Acupressure; Other: Listening Music; Other: Virtual Reality

INTERVENTIONS:
Other: Acupressure — Acupressure will be administered by a researcher who has completed the Acupressure application course at Ankara Başkent Personal Training Institutions and received their certificate. To determine the child's ability to assess the scale, they will be asked, "Is 8 bigger than 4?". Before the acupressure application, the child's area will be prepared in the blood collection room. Hands will be washed and warmed by rubbing before the acupressure application. Pressure will be applied for 1.5 minutes to point 4 of the large intestine (LI4), located on the radial side of the 2nd metacarpal bone, at the junction of the 1st and 2nd metacarpal bones, on the back of the hand. Then, the blood collection nurse will begin the blood collection procedure from the same arm. Pressure will continue for another 1.5 minutes while the blood collection procedure continues. In total, pressure will be applied to point LI4 for 3 minutes: 1.5 minutes before and 1.5 minutes during the procedure.
  Arms: Experimental Group
Other: Listening Music — Before the procedure, children will be given brief and understandable information, and if possible, calming and age-appropriate music will be chosen according to their musical preferences. The music will start 1-2 minutes before the procedure begins and continue through headphones or speakers during blood collection to distract the child's attention from the needle; it will also be played for another 1-2 minutes afterward to help the child relax and complete the procedure as a positive experience. During this process, the children's pain, fear, and anxiety levels will be measured.
  Arms: Experimental Group
Other: Virtual Reality — In this study, children will be shown cartoons via virtual reality glasses during blood collection. For both boys and girls, the content options will be the 360-degree virtual reality cartoon "Ice Age," chosen by experts in child development and psychology to be age and gender-appropriate. The suitability of "Ice Age" for children was evaluated by five academics specializing in child health, and all experts deemed it appropriate. Children will begin watching the cartoon via VR approximately 3 minutes before blood collection and will continue watching until the procedure is complete.
  Arms: Experimental Group

SUMMARY:
This study aims to evaluate the effects of acupressure, music listening, and virtual reality applications, which appeal to the senses of touch, hearing, and sight during blood sampling, on pain, fear, and anxiety levels in children.

DETAILED DESCRIPTION:
Two hundred volunteer children aged 5-10 coming for blood collection will be randomly divided into four groups: acupressure, virtual reality, Listening music and control group. Children will be assessed before, during, and after the procedure. Pain related to blood collection will be assessed with the Wong-Baker Faces Pain Scale, fear will be assessed with the Child Fear Scale and anxiety will be assessed with the Child Anxiety Scale - State. In addition, children's demographic data will be recorded in the Information Form.

ELIGIBILITY:
Inclusion Criteria:

Being between 5-10 years old Being healthy (no chronic disease diagnosis) Both child and parent agree to participate in the study Being able to communicate in Turkish Taking a blood sample in a single session Having no visual, auditory, or speech impairments, Being open to communication Being accompanied by a parent

Exclusion Criteria:

Having an allergy to any substance Having a chronic illness (Type 1 diabetes, etc.) Having upper respiratory tract diseases such as asthma, rhinitis, pharyngitis Having an obstructive condition in the nasal passages for any reason Having vision or hearing loss Having any neuropathological problem Having complaints of vomiting, nausea, or pain Having recently used sedatives, anesthetics, or analgesics Having a chronic illness Having visual-auditory and speech impairments History of sedative, analgesic, or narcotic substance use within 24 hours prior to admission

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
1. Patient Identification Form | Baseline
  The form consists of a total of 7 questions covering the child's age, gender, previous hospital experience (if any), number of hospitalizations, whether their parents prepared them for blood tests beforehand, their experience with blood tests in the last six months, and their reactions to the blood test procedure.
Wong Baker Face Pain Scale | Baseline and up to 4 weeks
  Children between the ages of three and eight can express many pain areas and their severity. In this study, the Wong-Baker Pain Inventory will be used in combination with the Visual Analog Scale, since face scales are more appropriate. The Wong Baker Face Pain Scale was developed by Donna Wong and Connie Moran Baker in 1981. The scale is suitable for children between the ages of three and eighteen. The scale includes facial expressions that the child can enjoy and enjoy. For this reason, it has been stated that it gives more accurate results. The scale has scores of "0", "2", "4", "6", "8", and "10". A score of "0" indicates no pain and a score of "10" indicates the highest pain. This scale does not have a Cronbach's alpha score. It has been reported that reliability studies have not been conducted on such scales.
3. Child Fear Scale | Baseline and up to 4 weeks
  The Turkish validity of this scale, developed by McMurtry and colleagues, was done by Gerçeker and colleagues. The changes in the facial muscles of the frightened expression were drawn by a graphic artist from a photograph of a frightened face. It can be used by the parent, child or researcher to scale the child's fear. The scale, which has facial expressions scored from 0 to 4, is shown to the child. A score of 4 indicates that the child is very frightened, and a score of 0 indicates that the child is not frightened. It is accepted that a score of "0" indicates a neutral expression (no fear), a score of "1" indicates a very low level of fear, a score of "2" indicates a little fear, a score of "3" indicates a greater level of fear, and a score of 4 indicates that the level of fear is at the highest level. This scale can be used to measure fear before and during the procedure.
4. The Child Anxiety Scale-State (CAS-S) | Baseline and up to 4 weeks
  Developed by Ersig et al. in 2013, the Child Anxiety Scale-State measures situational anxiety in children aged 4-10 years. Its validity was established by Gerçeker et al. in 2017. The CAS-S (State) is designed as a thermometer. At the bottom is a bulb, and horizontal lines extend upwards. Each horizontal line represents a score, and the thermometer has 10 points. The bulb at the bottom represents 0 points, indicating no anxiety. As the lines rise, anxiety increases. The peak, worth 10 points, represents the highest level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze AKAY, 1, Principal Investigator — Artvin Coruh University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oluc T, Sarialioglu A. The effect of a hand puppet-based therapeutic play for preschool children on the fear and pain associated with blood collection procedure. J Pediatr Nurs. 2023 Sep-Oct;72:e80-e86. doi: 10.1016/j.pedn.2023.06.012. Epub 2023 Jun 15. PMID 37330277
- See also: Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/37330277/